CLINICAL TRIAL: NCT05192057
Title: A Randomized Controlled Trial on Hypertonic Saline Inhalation in Patients With Nodular-bronchiectatic Mycobacterium Avium Complex Pulmonary Disease
Brief Title: Hypertonic Saline Inhalation for Mycobacterium Avium Complex Pulmonary Disease
Acronym: SALINE
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Radboud University Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: KGx60
Record Dates: First submitted 2021-12-29; First posted 2022-01-14 (Actual); Last update posted 2025-06-26 (Actual); Status verified 2025-06

CONDITIONS: Nontuberculous Mycobacterial Lung Disease; Mycobacterium Avium Complex
MeSH Terms: conditions — Mycobacterium avium-intracellulare Infection

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Hypertonic Saline inhalation (Experimental): Participants randomized to the Hypertonic Saline inhalation arm will be prescribed a nebulizer for Hypertonic Saline Inhalation (5ml, 5.8%) two times a day for 12 weeks. Participants will also receive best supportive care for 12 weeks (see below).
  Interventions: Device: Hypertonic Saline inhalation
- Best supportive care (No Intervention): Participants randomized to the best supportive care arm will receive standard of care including management of predisposing (lung) disease, guidance in smoking cessation, respiratory physiotherapy (e.g. airway clearance), nutritional guidance, but no antimycobacterial treatment.

INTERVENTIONS:
Device: Hypertonic Saline inhalation — Hypertonic Saline inhalation is thought to increase mucociliary clearance of the airways
  Arms: Hypertonic Saline inhalation

SUMMARY:
The SALINE trial will investigate the effect of Hypertonic Saline inhalation plus best supportive care on burden of symptoms, clearance of mycobacteria and functional capacities in participants with Mycobacterium avium complex lung disease and compare the effect to treatment with best supportive care alone.

DETAILED DESCRIPTION:
The treatment of Mycobacterium avium complex (MAC) lung disease consists of best supportive care, often accompanied by long-lasting multi-drug antibiotic regimens. Two major radiologic patterns exist: nodular-bronchiectatic and fibrocavitary disease, characterized by slow and rapid progression of disease, respectively.

SALINE is an open-label, randomized, two-arm controlled study that investigates the effect of Hypertonic Saline inhalation (HSi) plus best supportive care versus best supportive care alone for 12 weeks in participants with nodular-bronchiectatic MAC lung disease. The investigators hypothesize that HSi added to best supportive care will improve health-related quality of life and reduce mycobacterial load more than best supportive care alone Participants will be randomized 1:1 to a study arm. Best supportive care comprises of management of a predisposing (lung) condition, guidance in smoking cessation, respiratory physiotherapy (e.g. airway clearance) and nutritional guidance. HSi will be administered two times daily. Antibacterial therapy against other bacterial infections and inhaled corticosteroids are allowed during the study period.

ELIGIBILITY:
Inclusion Criteria:

* International guideline criteria for nodular-bronchiectatic MAC lung disease, i.e. symptomatic, nodular bronchiectatic lesions seen on thorax radiography and ≥2 positive cultures of the same MAC species or one positive culture from a bronchoalveolar lavage;
* ≥1 positive MAC sputum cultures must be collected in the previous 4 months;
* Signed and dated patient informed consent.

Exclusion Criteria:

* Fibrocavitary MAC lung disease;
* Antimycobacterial treatment in the last 6 months;
* Previous MAC lung disease treatment failure, defined as persistent culture positivity despite >6 months of guideline-recommended treatment;
* Current clinical relevant asthma or otherwise bronchial hyperresponsiveness that is judged to be a contra-indication for HSi.
* Current HSi use
* Former adverse reaction to HSi (note: former HSi use that was stopped due to a lack of clinical improvement is not an exclusion criterium);
* Hypertonic saline intolerability during the screening test inhalation
* Diagnosis of HIV;
* Diagnosis of Cystic fibrosis (CF);
* Active pulmonary malignancy (primary or metastatic) or any other malignancy requiring chemotherapy or radiotherapy within 6 months before screening or anticipated during the study period;
* Active pulmonary tuberculosis, fungal or nocardial disease requiring treatment
* Current use of chronic systemic corticosteroids at doses of 15 mg/day for more than 3 months
* Prior lung or other solid organ transplant
* Known or suspected current drug or alcohol abuse, that is, in the opinion of the Investigator, sufficient to compromise the safety or cooperation of the patient.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2022-05-20 (Actual); Primary Completion 2026-10-01 (Estimated); Study Completion 2026-10-01 (Estimated)

PRIMARY OUTCOMES:
Change in health-related quality of life | 12 weeks
  Measured by the Quality of Life - Bronchiectasis (QOL-B) with NTM module questionnaire at baseline, after 4, 8 and 12 weeks. The QOL-B asks the participant to subjectively rank their symptoms using a 4 scale base ranging from "a lot of difficulty" to "no difficulty", "always" to "never", "completely true" to "not at all true" and "a lot" to "not at all" for 8 domains: physical/role/emotional/social functioning, vitality, treatment burden, health perception and respiratory symptoms. The NTM-module also asks participants to subjectively rank eating problems, body image, digestive symptoms, and NTM symptoms on a 4 scale base.
Change in health-related quality of life | 12 weeks
  Measured by the PROMIS Fatigue 7a short form at baseline, after 4, 8 and 12 weeks. This questionnaire assesses self-reported fatigue over the past seven days on a 5 scale base ranging from never (1) to always (5). The lowest possible raw score (indicating the highest subjective level of fatigue) is 7; and the highest possible raw score (indicating the lowest subjective level of fatigue) is 35.

SECONDARY OUTCOMES:
Sputum culture conversion | 12 weeks
  A conversion from positive sputum cultures at baseline to negative sputum cultures after study treatment, defined by two or more negative sputum cultures sampled a week apart.
Change in semi-quantitative culture results | 12 weeks
  Change in acid fast bacilli (AFB) smear determined by auramine staining
Change in semi-quantitative culture results | 12 weeks
  Change in sputum culture time-to-positivity
(Serious) Adverse Events as assessed by CTCAE v5.0 | 12 weeks
  Number and severity of (serious) Adverse Events as assessed by CTCAE
Treatment failure | 12 weeks
  Progression of disease that requires the start of antimycobacterial treatment as per the treating physician's discretion.
Change in pulmonary function parameters | 12 weeks
  Forced expiratory volume in 1 second (FEV1; L), Forced Vital Capacity (FVC; L), Inspiratory Capacity (IC; L), Functional Residual Volume (FRC; L) and Total Lung Capacity (TLC; L).
Change in pulmonary function parameters | 12 weeks
  Tiffeneau index (FEV1/FVC; %)
Change in physical function capacity | 12 weeks
  Change in 6-Minute Walking Distance (6MWD).
Change in inflammatory serum biomarkers | 12 weeks
  Change in C-reactive protein (CRP).
Change in inflammatory serum biomarkers | 12 weeks
  Erythrocyte Sedimentation Rate (ERS)
Change in inflammatory serum biomarkers | 12 weeks
  White blood cell count.
Therapy adherence | 12 weeks
  Self-reported therapy adherence expressed as percentage taken of total HSi administrations.
Change in self-reported health status | 12 weeks
  Change in the Nijmegen Clinical Screening Instrument (NCSI) from baseline to 12 weeks. The NCSI evaluates clinical, social and emotional self-reported measures, serves as a tool for an individualized treatment plan and can be repeated regularly to monitor the treatment effect

CONTACTS AND LOCATIONS:
Locations (1):
- Radboud University Medical Center, Nijmegen, Netherlands